CLINICAL TRIAL: NCT04811235
Title: "OMNI-SCI" Trial - "Optical Monitoring With Near-Infrared Spectroscopy for Spinal Cord Injury" Trial
Brief Title: Optical Monitoring With Near-Infrared Spectroscopy for Spinal Cord Injury Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Brian Kwon, MD, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: H20-01259.
Record Dates: First submitted 2021-03-15; First posted 2021-03-23 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Acute Spinal Cord Injury; Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): NIRS monitoring of spinal cord oxygenation and hemodynamics
  Interventions: Device: Near Infra-Red Spectroscopy (NIRS) Sensor

INTERVENTIONS:
Device: Near Infra-Red Spectroscopy (NIRS) Sensor — The NIRS sensor is laid on top of the dura, at the site of the SCI, and emits near-infrared light signals into the cord to measure tissue oxygenation and tissue hemodynamics in real-time.

SUMMARY:
The study involves the 'first-in-human' evaluation of a novel optical sensor which uses near-infrared spectroscopy (NIRS) technology to assess oxygenation and hemodynamics of the injured spinal cord. The NIRS sensor is laid on top of the dura, at the site of the SCI, and emits near-infrared light signals into the cord to measure tissue oxygenation and tissue hemodynamics in real-time. Our testing of this novel NIRS sensor in patients with acute SCI represents the first step in translating this technology for human use.

DETAILED DESCRIPTION:
This single-center, prospective observational study will enroll 10 patients admitted to Vancouver General Hospital (VGH) for treatment of an acute traumatic spine injury.

Promising preclinical data demonstrates that the oxygenation and hemodynamic measures of our Near Infra-Red Spectroscopy (NIRS) system closely match the invasive intraparenchymal measures obtained within the injured spinal cord. Further, the NIRS sensor is responsive and reflective of systemic hemodynamic changes. This clinical protocol represents the first application of this novel NIRS sensor in human SCI. Following operative decompression of the spinal cord via a posterior approach, the NIRS sensor will be placed over the dura for 7 days to monitor spinal cord oxygenation and tissue hemodynamics. Patients will be followed for 6 months and data collection for safety, feasibly and efficacy of the NIRS System.

The specific aims of this project are to:

1. Establish the safety, feasibility, and efficacy of our NIRS system in monitoring tissue oxygenation and hemodynamics of the injured spinal cord in human participants.
2. Complete the technical refinement of the NIRS system utilizing an iterative process guided by participant recruitment and data accrual during the trial.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 17 years or older
* Spinal injury between bony levels C3 and L1 inclusive
* Motor complete acute traumatic SCI (AIS A or B) or motor incomplete SCI (AIS C) with a total lower extremity motor score of less than 5
* Blunt (non-penetrating) SCI requiring posterior laminectomy with stabilization/fusion surgery within 72 hours of injury
* Able to communicate in English and provide informed consent

Exclusion Criteria:

* Isolated radiculopathy or cauda equina injury
* Spinal cord impairment secondary to tumour, infection, epidural bleeding, or ischemia (in
* Any condition or injury (e.g. Morel-Lavellee lesion) that would interfere with the application or readings of the NIRS sensor
* Associated traumatic condition that would interfere with the informed consent process or outcome assessments (e.g. traumatic brain injury, pelvic, abdominal, or thoracic injuries)
* Any other medical condition that, in the investigator's opinion, would render the protocol procedures dangerous
* Female patients who are pregnant

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-09-24 (Actual); Primary Completion 2024-06-02 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility Assessment - Overall | Day 7
  Study specific questionnaire will collected data on the the ease of sensor application, NIRS monitoring and sensor removal is recorded with this form. Series of questions requiring the assessment of the NIRS system using yes/no and 10-point scoring scale
Feasibility Assessment: Sensor Application | Day 1
  Study specific form will be used record data associated with application of the NIRS sensor, such as the laminectomy and instrumentation data, location of the sensor and ease of application (score out of 10).
Feasibility Assessment: Sensor Removal | Day 7
  Study specific form will be used to record the condition of the sensor and participants' experience (score out of 10) at the time of sensor removal

OTHER OUTCOMES:
Safety Assessment - Neurologic Function | 6 Month
  Neurologic function will be assessed using the International Standards for Neurologic Classification of Spinal Cord Injury (ISNCSCI) to determine if the application, 7-day placement, or removal of the NIRS sensor is associated with any deterioration in spinal cord function.
Safety Assessment - Wound Assessment | Day 7
  The externalization of a foreign body may lead to an increased risk of surgical site infection. Any incidence of wound infection will be monitored and document on a wound assessment form.
Safety Assessment - Adverse Events | 6 Months
  The incidence of AEs in the acute SCI patient population is significant. For the purposes of this study, and in keeping with standard of care on the Acute Spine Unit at study site, all AEs will be recorded utilizing the Spine Adverse Event (SAVES) form, a well-established system for prospectively documenting AEs in spine patients

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kwon, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada